CLINICAL TRIAL: NCT06343948
Title: A Phase III Randomized Controlled Clinical Study Comparing BL-B01D1 With Chemotherapy of Physician's Choice in Patients With Unresectable Locally Advanced, Recurrent, or Metastatic HR+HER2- Breast Cancer After Failure of at Least One Prior Line of Chemotherapy
Brief Title: A Study Comparing BL-B01D1 With Chemotherapy of Physician's Choice in Patients With Unresectable Locally Advanced, Recurrent, or Metastatic HR+HER2- Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-306
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: HR+HER2- Breast Cancer
MeSH Terms: interventions — eribulin; Vinorelbine; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-B01D1 (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1
- Eribulin or Vinorelbine or Gemcitabine or Capecitabine (Experimental): Participants receive Eribulin or Vinorelbine or Gemcitabine or Capecitabine in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Eribulin; Drug: Vinorelbine; Drug: Gemcitabine; Drug: Capecitabine

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
  Arms: BL-B01D1
Drug: Eribulin — Administration by intravenous bolus for a cycle of 3 weeks.
  Arms: Eribulin or Vinorelbine or Gemcitabine or Capecitabine
Drug: Vinorelbine — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Eribulin or Vinorelbine or Gemcitabine or Capecitabine
Drug: Gemcitabine — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Eribulin or Vinorelbine or Gemcitabine or Capecitabine
Drug: Capecitabine — Oral administration for a cycle of 3 weeks.
  Arms: Eribulin or Vinorelbine or Gemcitabine or Capecitabine

SUMMARY:
This trial is a registered phase III, randomized, open-label, multicenter study to evaluate the efficacy and safety of BL-B01D1 in patients with unresectable locally advanced, recurrent, or metastatic HR+HER2- breast cancer after failure of at least one prior line of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. No gender limit;
3. Age ≥18 years old;
4. expected survival time ≥3 months;
5. Patients with unresectable locally advanced, recurrent metastatic HR+HER2- breast cancer;
6. The subjects had received 1-2 lines of chemotherapy regimens in the unresectable locally advanced recurrence or metastasis stage, and had been treated with endocrine, CDK4/6 inhibitors, and taxanes;
7. Documented radiographic disease progression;
8. Consent to provide archival tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 3 years;
9. Must have at least one measurable lesion according to RECIST v1.1 definition;
10. ECOG score 0 or 1;
11. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
12. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
13. No blood transfusion, no use of cell growth factors and/or platelet raising drugs within 14 days before screening, and the organ function level must meet the requirements;
14. Urine protein ≤2+ or < 1000mg/24h;
15. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, serum pregnancy must be negative, and it must be non-lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Prior receipt of an ADC drug with a topoisomerase I inhibitor as a toxin;
2. Prior receipt of an ADC or antibody drug targeting EGFR and/or HER3;
3. Chemotherapy, biological therapy, immunotherapy, etc., have been used within 4 weeks or 5 half-lives before the first dose, small molecule targeted therapy has been used within 5 days, palliative radiotherapy, modern Chinese medicine preparations approved by NMPA for anti-tumor therapy, etc., have been used within 2 weeks;
4. anthracycline equivalent cumulative dose of adriamycin > 360 mg/m2;
5. History of severe cardiovascular or cerebrovascular disease;
6. Unstable deep vein thrombosis, arterial thrombosis, and pulmonary embolism requiring medical intervention within 6 months before screening; Infusion-related thrombosis was excluded;
7. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
8. Other malignant tumors diagnosed within 3 years before the first dose;
9. Hypertension poorly controlled by two antihypertensive drugs; Patients with poor glycemic control;
10. A history of interstitial lung disease (ILD) requiring steroid therapy, current ILD or grade ≥2 radiation pneumonitis, or suspicion of such disease on imaging during screening;
11. Complicated pulmonary diseases leading to clinically severe respiratory function impairment;
12. Patients with active central nervous system metastases;
13. Patients with massive or symptomatic effusions or poorly controlled effusions;
14. Imaging examination showed that the tumor had invaded or wrapped around the large blood vessels in the abdomen, chest, neck, and pharynx;
15. Severe infection within 4 weeks before randomization; Evidence of pulmonary infection or active pulmonary inflammation within 2 weeks before randomization;
16. Was receiving &gt before randomization; Long-term systemic corticosteroid therapy with 10mg/ day prednisone or equivalent anti-inflammatory active drugs or any form of immunosuppressive therapy;
17. Severe unhealed wound, ulcer, or fracture within 4 weeks before signing the informed consent;
18. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
19. Patients with inflammatory bowel disease, extensive bowel resection history, immune enteritis history, intestinal obstruction or chronic diarrhea;
20. Have a history of allergy to recombinant humanized antibodies or to BL-B01D1 and any excipients; A history of autologous or allogeneic stem cell transplantation;
21. Human immunodeficiency virus antibody positive, active hepatitis B virus infection or hepatitis C virus infection;
22. A history of severe neurological or psychiatric illness;
23. Received other unmarketed investigational drug or treatment within 4 weeks before the first dose; A live vaccine dose within 28 days before the planned dose or the first dose;
24. Any complications or other circumstances deemed by the investigator to preclude participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China